CLINICAL TRIAL: NCT03366688
Title: A Randomized, Double Blind, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics/Pharmacodynamics of IBI306 in Healthy Subjects.
Brief Title: Single Ascending Dose Study of PCSK-9 Inhibitor (IBI306) in Healthy Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CIBI306A101
Record Dates: First submitted 2017-11-27; First posted 2017-12-08 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI306 (Active Comparator): Subcutaneous or intravenous injection of a single dose of IBI306, dose level according to ascending dose design
  Interventions: Drug: IBI306
- placebo (Placebo Comparator): Subcutaneous or intravenous injection of a single dose of placebo, dose level according to ascending dose design
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: IBI306 — Cohort 1: 25 mg Subcutaneous(SC) (this cohort is open label without placebo); Cohort 2: 75 mg SC; Cohort 3: 150 mg SC; Cohort 4: 75 mg IV; Cohort 5: 300 mg SC; Cohort 6: 450 mg SC; Cohort 7: 600 mg SC; Cohort 8: 450 mg IV.
  Arms: IBI306
Drug: placebo — Cohort 2: 75 mg SC; Cohort 3: 150 mg SC; Cohort 4: 75 mg IV; Cohort 5: 300 mg SC; Cohort 6: 450 mg SC; Cohort 7: 600 mg SC; Cohort 8: 450 mg IV.
  Arms: placebo

SUMMARY:
IBI306 is a fully human monoclonal antibody that binds proprotein convertase substilisin/kexin type 9 (PCSK9), preventing its interaction with the low-density lipoprotein cholesterol receptor (LDL-R) and thereby restoring LDL-R recycling and low-density lipoprotein cholesterol（LDL-C）uptake. This is a randomized, double-blind, placebo-controlled,single ascending dose study to evaluate the safety, tolerability, pharmacokinetics/pharmacodynamics and immunogenicity of IBI306 in healthy adults.

DETAILED DESCRIPTION:
Ascending dose design includes 6 dose levels （25 mg, 75 mg, 150 mg, 300 mg, 450 mg and 600 mg). Tolerance and safety data up to 14 days after dosing from all subjects of the previous cohort will be reviewed before proceeding to the next dose. Total duration of the study per subject is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chinese healthy men or women aged 18 to 55 years old at screening (inclusive）;
* Serum LDL-C concentration between 1.8 mmol/L and 4.9 mmol/L (inclusive）at screening;
* Body mass index between 19 and 28 kg/m2 (inclusive);
* Willing to maintain the current regular diet and physical activity;
* Female subjects and male subject's partner who could become pregnant should take effective contraceptions during the treatment period and 6 months after dosing;
* Without any medical history of serious diseases;
* Willing to comply with protocol required visit schedule and visit requirements and provide written informed consent.

Exclusion Criteria:

* Breast-feeding or pregnant women;
* History of allergic reaction;
* Previously received any anti-PCSK-9 treatment;
* Vital signs, physical examination, clinical laboratory test, 12-lead ECG, and chest X-ray are abnormal with clinical significance;
* Not willing to stop intense physical activities (such as weight lifting or long-distance running) before 72 hours of the scheduled visits;
* Any hospitalization within one month before screening, or major surgery within six months before screening, or any other unstable medical condition;
* Received an investigational chemical agent within 30 days before dosing；
* Received an investigational biological agent within 90 days before dosing；
* Use of medications including over-the-counter medication within 14 days or less than 5 half-lifes of the agent;
* Use of herb,vitamins or nutraceutical in order to alter serum lipids;
* Positive screen of hepatitis B surface antigen, hepatitis C virus, human immunodeficiency virus or syphilis infection at screening；
* History or clinical evidence of alcohol or drugs of abuse within 12 months before screening;
* With any consumption of alcohol and caffeinated beverages within 72 hours prior to and during the trial;
* Blood donations or blood loss 200 ml and more within 2 months before screening;
* History of organ transplantation or malignant tumor;
* Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events（AEs) as assessed by the criteria of National Institute on Aging | up to 12 weeks

SECONDARY OUTCOMES:
The area under the curve (AUC) of serum concentration of the drug after the administration | up to 12 weeks
Maximum concentration (Cmax) of the drug after the administration | up to 12 weeks
Time at which maximum concentration (Tmax) occurs for the drug after the administration | up to 12 weeks
The half-life (t1/2) of drug after the administration | up to 12 weeks
Assessment of serum concentrations of PCSK-9 | up to 12 weeks
Change from baseline in lipid parameters | up to 12 weeks
Number of participants with anti-drug antibodies or neutralizing antibodies | up to 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the study protocol with any amendments and statistical analysis plan. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants.
Supporting Information: Study Protocol, SAP